CLINICAL TRIAL: NCT00586118
Title: Inhalative Sedation in ICU With Sevoflurane Via Anaesthetic Conserving Device Compared to Propofol
Status: Completed | Type: Observational
Sponsor: Klinikum Ludwigshafen (Other)
Collaborators: Universitätsmedizin Mannheim (Other)
Responsible Party: Klinkum Ludwigshafen, Department of Anaesthesiology and Intensive Care, Dr. K. D. Röhm, Klinikum Ludwigshafen, Dep. of Anaesthesiology
Other Study IDs: ANA06104; ANA06104
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Recovery From Sedation; Sevoflurane Consumption; Renal Function; Hepatic Function; Cardioprotection
Keywords: Sedation; Volatile anaesthetic; Sevoflurane; Propofol; Recovery
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1-Sevo: Sevoflurane/ACD group (n=60)
  Interventions: Drug: Sevoflurane
- 2-Propofol: Propofol group (n=60)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane sedation, 0.5-1 Vol%, continuously via syringe pump, up to 72 hours in ICU
  Other Names: Sevorane (Abbott GmbH, Wiesbaden, Germany)
  Groups: 1-Sevo
Drug: Propofol — Propofol, 1.5-3 mg/kgBW/h, continuously via syringe pump, up to 72 hours
  Other Names: disoprivan
  Groups: 2-Propofol

SUMMARY:
The evaluation of the presented study will work on the practicability of inhalative sedation on the ICU, potential benefits and limitations of the ACD system in a postoperative sedated patient population in comparison to a standard intravenous sedation regimen with propofol, and focus on renal and hepatic function, cardioprotection and pharmacoeconomics

DETAILED DESCRIPTION:
A goal-oriented sedation complies the ability to sedate the patient as deeply as necessary, and allow a modern ventilation regimen with early spontaneous breathing and a pain-free cooperative patient. The ideal sedative agent - with a short duration of action, predictable wake-up times, low drug toxicity, haemodynamic stability and less side effects, and a rational pharmacoeconomic impact nowadays - has still to be found. Inhalative anaesthetics show these properties, but until the introduction of AnaConDa© (Anesthetic Conserving Device, ACD) in 2005, the use of volatile anaesthetics on the intensive care unit (ICU) required specific evaporating devices or scavenging systems. The ACD, a modified heat- moisture filter, is connected to the breathing circuit of conventional ICU ventilators and a syringe pump delivers the volatile anaesthetic to the ACD where it is vaporized through a rod. Most of the exhaled gas is absorbed in a charcoal filter's membrane and reflected to the patient in the following inspiration. Randomised, controlled and comparative studies to the use of volatile anaesthetics in ICU via this innovative device are still missing. Isoflurane has been studied in small patient populations and in comparison to midazolam, while Sevoflurane - a newer volatile agent with short action, brief elimination time, and low hepatic biodegradation - has only been studied intraoperatively and in short-term sedation. This is the first prospective, randomised, clinical study on the feasibility of sevoflurane via the ACD for sedation in ICU patients until 72 hours in comparison to a standard intravenous sedation with propofol. The investigation will work on potential benefits and limitations of the use of volatile agents on the ICU, the quality of sedation (Richmond Agitation Sedation Scale, BIS), infusion rate stability of sevoflurane and respiratory parameters, short-term recovery (time from discontinuation of infusion until following verbal commands and extubation), haemodynamics, renal and hepatic function and adverse side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* elective operative procedure, and indication for admission to the ICU for postoperative sedation
* ASA I-III
* weight 50-120 kg
* Haemoglobin > 10 g/dl
* ability and acceptance to agree to the study participation

Exclusion Criteria:

* malignant hyperthermia
* muscle diseases or weakness
* liver insufficiency (ASAT, ALAT > 40 U/min)
* pancreas insufficiency
* emergencies
* women in child bearing age and missing negative pregnancy test, pregnancy or lactation
* diseases from the central nervous system (such as M. Parkinson and multiple sclerosis)
* increased intracranial pressure, head trauma
* pre-existing delirium, agitation and psychiatric derangements
* alcohol and drug abuse (including opioid abuse)
* allergy to any of the study agents
* refusal from the patient to participate in the study
* participation in another study project.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 patients, scheduled for elective major surgery and postoperative admission to the ICU, are screened the day before surgery for potential in- and exclusion criteria.
Enrollment: 120 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Extubation time | Termination of sedation to extubation

SECONDARY OUTCOMES:
Consumption of anaesthetics | until discharge from hospital
Renal function | until discharge from hospital
Hepatic function | until discharge from hospital
Cardioprotection | until discharge from hospital
Costs | until discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin D. Röhm, Dr. med., Principal Investigator — Klinikum Ludwigshafen, Department of Anaesthesiology, Ludwigshafen, Germany

REFERENCES:
- [Background] Sackey PV, Martling CR, Nise G, Radell PJ. Ambient isoflurane pollution and isoflurane consumption during intensive care unit sedation with the Anesthetic Conserving Device. Crit Care Med. 2005 Mar;33(3):585-90. doi: 10.1097/01.ccm.0000156294.92415.e2. PMID 15753751
- [Background] Sackey PV, Martling CR, Granath F, Radell PJ. Prolonged isoflurane sedation of intensive care unit patients with the Anesthetic Conserving Device. Crit Care Med. 2004 Nov;32(11):2241-6. doi: 10.1097/01.ccm.0000145951.76082.77. PMID 15640636
- [Background] Berton J, Sargentini C, Nguyen JL, Belii A, Beydon L. AnaConDa reflection filter: bench and patient evaluation of safety and volatile anesthetic conservation. Anesth Analg. 2007 Jan;104(1):130-4. doi: 10.1213/01.ane.0000248221.44383.43. PMID 17179257